CLINICAL TRIAL: NCT00171834
Title: An Open Label, Phase I/II Dose Escalating Study Evaluating the Safety and Efficacy of EPO906, qw3, in Patients With Non-small Cell Lung Cancer.
Brief Title: Dose Escalating Study of the Safety and Efficacy of Patupilone, q3w, in Patients With Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEPO906A2209; NCT00088127 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2011-07-07 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: EPO; EPO906; Brain metastasis; Lung cancer; Lung metastasis; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms; Lung Neoplasms | interventions — epothilone B

INTERVENTIONS:
Drug: Patupilone — Patupilone (2.5 mg/mL) was supplied as a clear, colorless concentrate for solution for infusion in glass vials containing 5 mg/2 mL in Phase I and 10 mg/4 mL in Phase II part of the study. Patupilone was administered as a single intravenous (i.v.) infusion over 5 to 10 minutes (Amendment 1) till Amendment 2 and over 10 to 20 minutes (Amendment 2) till the completion of Phase I part of the study. Patupilone was administered as a single i.v. infusion over 20 minutes (Amendment 4), once every 3 weeks in Phase II part of the study.
  Other Names: EPO906; Epothilone B

SUMMARY:
The study objective is to evaluate the maximum tolerated dose, safety and efficacy of patupilone in patients with NSCLC who have progressed after prior chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologic or cytologic confirmation of unresectable locally advanced or metastatic NSCLC (stage IIIB with pleural effusion only / stage IV) documented before first line therapy.
* Prior treatment with a platinum-containing regimen
* Age ≥18 years.
* Performance status of 0-1 on the WHO scale.
* Life expectancy of ≥3 months.
* NSCLC patients should have at least one measurable lesion as defined by modified RECIST criteria. If the patient has had previous radiation to the marker lesion(s), the lesion must have demonstrated progression since the radiation.
* NSCLC patients with controlled brain metastases are eligible to be enrolled in the brain metastases cohort at the MTD. "Controlled brain metastases" patients are defined as patients who are neurologically stable, i.e. have not experienced an increase in dose of steroidal or anticonvulsive therapy for at least 14 days prior to study entry.
* Patients with brain metastases must be verified to have metastases secondary to NSCLC based on histology of primary and by temporal sequence of events (note: these patients are eligible even if lung disease is quiescent).
* Patients with brain metastases must show evidence of residual disease or progression of disease since prior radiological or surgical therapy.
* Patients with brain metastases should have at least one bidimensionally measurable intracranial lesion of minimum diameter 2 cm. Multifocal disease is permitted, but the eligibility of BM patients presenting with more than 6 intracranial lesions should be discussed with Novartis prior to enrolling the patient.
* Patients with adequate hematologic parameters:
* ANC ≥1.5 x 10^9/L;
* Hb ≥9.0 g/dL,
* Platelet count ≥100 x 10^9/L (untransfused).
* Demonstrate the following blood chemistry laboratory values:
* total bilirubin ≤ 1.5 x ULN;
* AST/ALT ≤ 2.5 X ULN; (≤ 5 x ULN if hepatic metastasis is present)
* alkaline phosphatase ≤ 2.5 x ULN; (≤ 5 x ULN if hepatic and/or bone metastasis are present)
* serum creatinine < 2 x ULN.
* Female patients must have a negative serum pregnancy test at screening. (Not applicable to patients with bilateral oophorectomy and/or hysterectomy or to those patients who are postmenopausal).
* All patients of reproductive potential must agree to use an effective method of contraception during the study and three months following termination of treatment.
* All patients must use a barrier method for contraception for sexual intercourse or avoid this for the first 5 days after patupilone infusion.
* Written informed consent must be obtained.

Exclusion Criteria:

* Patients who have received more than one prior chemotherapy regimen or any other systemic antineoplastic treatment including immunotherapy.
* Patients who have received any investigational compound within the past 28 days or who are planning to receive other investigational drugs while participating in the study.
* Patients with brain metastases who have received any prior chemotherapy regimen or any other systemic antineoplastic treatment for brain metastases.
* Patients with brain metastases who have experienced a dose increase of 25% or more above previous dose, in concomitant steroidal or anticonvulsive therapy within 14 days prior to study entry.
* Patients with brain metastases receiving steroidal or anticonvulsive therapy for whom a dose increase has been required within 14 days prior to start of study drug.
* Patients with brain metastases who have leptomeningeal disease.
* Patients with brain metastases who have extracranial metastases in more than two organs.
* Patients with any peripheral polyneuropathy > Grade 1.
* Patients with unresolved diarrhea > Grade 1.
* Patients receiving hematopoietic growth factors except erythropoietin (refer Section 3.4.4).
* Severe cardiac insufficiency (NYHA III or IV), with uncontrolled and/or unstable cardiac or coronary artery disease.
* Patients taking warfarin or other agents containing warfarin, with the exception of low dose warfarin (1 mg or less daily) administered prophylactically for maintenance of in-dwelling lines or ports.
* Patients who have not recovered fully from surgery for any cause, including brain metastases patients who have had a biopsy or surgical resection of the brain tumor within 2 weeks prior to starting study drug or who are not fully recovered from any prior biopsy or surgical resection.
* Patients who have received radiation therapy or chemotherapy within the last four weeks. Palliative radiotherapy of metastasis in extremities is allowed but such lesions cannot be used as tumor markers.
* Patients with the presence of active or suspected acute or chronic uncontrolled infection, including abscess or fistulae.
* Patients known to be HIV positive.
* History of another malignancy within 3 years prior to study entry, except curatively treated non-melanotic skin cancer or cervical cancer in situ.
* For patients enrolling in the brain metastases cohort, any of the following exclusions to MRI imaging:

Cardiac pacemaker Ferromagnetic metal implants other than those approved as safe for use in MRI scanners Claustrophobia Obesity (exceeding the limits of scanning equipment)

* Pregnant or lactating females.
* A history of noncompliance to medical regimens or inability or unwillingness to return for all scheduled visits.

Other protocol-dependent inclusion / exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2003-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (4):
  - Norton Healthcare/Hospital Inc, Louisville, Kentucky
  - Ellis Fisher Cancer Center, Columbia, Missouri
  - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Patupilone ≤7.0 mg/m^2 (Phase I); Patupilone 7.5-8.0 mg/m^2 (Phase I); Patupilone 8.5-9.5 mg/m^2 (Phase I); Patupilone 10.0-11.5 mg/m^2 (Phase I); Patupilone 12.0-13.0 mg/m^2 (Phase I): Patupilone was administered as a single i.v. infusion over 5 to 10 minutes (Amendment 1) until (Amendment 2) and over 10 to 20 minutes (Amendment 2) until the completion of Phase I part of the study.
- Patupilone 10 mg/m^2 (Phase II) NSCLC Cohort; Patupilone 10 mg/m^2 (Phase II) NSCLC w.BM Cohort: Patupilone was administered as a single i.v. infusion over 20 minutes (Amendment 4), once every 3 weeks.
Period: Overall Study
Arm/Group | Patupilone ≤7.0 mg/m^2 (Phase I) | Patupilone 7.5-8.0 mg/m^2 (Phase I) | Patupilone 8.5-9.5 mg/m^2 (Phase I) | Patupilone 10.0-11.5 mg/m^2 (Phase I) | Patupilone 12.0-13.0 mg/m^2 (Phase I) | Patupilone 10 mg/m^2 (Phase II) NSCLC Cohort | Patupilone 10 mg/m^2 (Phase II) NSCLC w.BM Cohort
Started | 6 | 12 | 12 | 12 | 8 | 35 | 4
Completed 6 Cycles of Treatment | 0 | 0 | 1 | 0 | 2 | 1 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 12 | 12 | 12 | 8 | 35 | 4
Not completed — Adverse Event | 2 | 1 | 3 | 2 | 2 | 15 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 1 | 1 | 1 | 0
Not completed — Death from study indication | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Disease Progression | 4 | 8 | 8 | 9 | 2 | 18 | 3
Not completed — Treatment Duration Completed | 0 | 0 | 1 | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patupilone ≤7.0 mg/m^2 (Phase I) | Patupilone 7.5-8.0 mg/m^2 (Phase I) | Patupilone 8.5-9.5 mg/m^2 (Phase I) | Patupilone 10.0-11.5 mg/m^2 (Phase I) | Patupilone 12.0-13.0 mg/m^2 (Phase I) | Patupilone 10 mg/m^2 (Phase II) NSCLC Cohort | Patupilone 10 mg/m^2 (Phase II) NSCLC w.BM Cohort | Total
Number analyzed (Participants) | 6 | 12 | 12 | 12 | 8 | 35 | 4 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (12.01) | 59.4 (8.98) | 57.8 (9.31) | 57.6 (9.07) | 56.3 (13.31) | 63.3 (8.04) | 60.5 (9.71) | 57.9 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 4 | 4 | 2 | 10 | 2 | 30
  Male | 3 | 7 | 8 | 8 | 6 | 25 | 2 | 59
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 6 | 12 | 11 | 12 | 8 | 35 | 4 | 88
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Best Overall Response-Phase I
Description: This was defined as the number of participants whose best overall response was CR or PR by RECIST. Per RECIST: CR, all detectable tumor has disappeared; PR, a >=30% decrease in the sum of the longest dimensions of the target lesions (TLs) taking as a reference the baseline sum, no worsening of non-TLs, and no new lesions; Progressive disease (PD), a >=20% increase in TLs, clearly worsening of non-TLs, or emergence of new lesions; Stable Disease (SD), small changes that do not meet previously given criteria.
Time Frame: Best achieved overall response according to RECIST from start of study until study discontinuation. Imaging was assessed every second cycle (ie. approximately every 6 weeks) until disease progression or discontinuation. Average 18 weeks
Population: Full Analysis Set (FAS) consisted of all patients who received at least one dose of patupilone. Analysis of the primary and all secondary efficacy endpoints was performed based on this population. According to the Intention to Treat (ITT) principle, patients were analyzed based on the treatment to which they were assigned at study entry.
Measure: Number; unit: Participants
Arm/Group | Patupilone ≤7.0 mg/m^2 (Phase I) | Patupilone 7.5-8.0 mg/m^2 (Phase I) | Patupilone 8.5-9.5 mg/m^2 (Phase I) | Patupilone 10.0-11.5 mg/m^2 (Phase I) | Patupilone 12.0-13.0 mg/m^2 (Phase I)
Number analyzed (Participants) | 6 | 12 | 12 | 12 | 8
Participants
  Complete Response (CR) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Partial Response (PR) | 0 (0) | 3 (25) | 1 (8.3) | 1 (8.3) | 0 (0)
  Stable Disease (SD) | 1 (16.7) | 2 (16.7) | 5 (41.7) | 4 (33.3) | 5 (62.5)
  Progressive Disease (PD) | 5 (83.3) | 4 (33.3) | 5 (41.7) | 6 (50.0) | 1 (12.5)
  Unknown | 0 (0) | 3 (25.0) | 1 (8.3) | 1 (8.3) | 2 (25.0)
  Best overall response (CR,PR) & the response rate | 0 (0) | 3 (25.0) | 1 (8.3) | 1 (8.3) | 0 (0)

2. Secondary Outcome: Overall Survival Time-Phase I and Phase II
Description: Overall survival (OS) time was measured from the start of study drug to the date of death due to any cause. If a patient was not known to have died, survival was censored at the date of last contact. Data was collected post treatment every 3 months until approximately 70% of patients have reached the survival endpoint (Phase I + Phase II).
Time Frame: From start of study drug to date of death due to any cause. Follow-up after treatment discontinuation approximately every 3 months until approximately 70% of participants have reached the survival endpoint. Average 9.75 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Patupilone (EPO906) Phase I | Patupilone (EPO906) Phase II
Number analyzed (Participants) | 50 | 35
Months | 9.2 [6.8 to 12.9] | 10.3 [6.0 to 13.6]

3. Secondary Outcome: Time to Progression (TTP)-Phase I and Phase II
Description: Time to progression was measured from the start of study drug to the date of first documented disease progression by RECIST, discontinuation due to disease progression, or death from underlying cancer, whichever event occurred first. If a patient had not progressed by RECIST, discontinued due to disease progression, or died from underlying cancer, TTP was censored at the time of last adequate tumor assessment. However, if a patient took any new cancer therapy prior to PD or death, then TTP was censored at the date of last adequate tumor assessment prior to the start date of new cancer therapy.
Time Frame: From baseline, then every second cycle (i.e. approximately every 6 weeks), until disease progression or discontinuation from study. Average 18 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Patupilone (EPO906) Phase I | Patupilone (EPO906) Phase II
Number analyzed (Participants) | 50 | 35
Months | 2.1 [0.8 to 3.5] | 2.1 [1.9 to 3.7]

4. Primary Outcome: Phase I: Number of Total Dose-limiting Toxicity (DLT) During Dose Escalation to Determine Maximum Tolerated Dose (MTD)
Description: The MTD was defined as the highest dose of patupilone administered every three weeks (q3w) where not more than one out of six patients experienced a DLT using a standard 3+3 design. Dose escalation started at 6.5 mg/m^2 until MTD in steps of 0.5 mg/m^2 until 12 mg/m^2, then in steps of 1 mg/m^2 till 13.0 mg/m^2. DLTs were assessed during cycle 1. During this time frame, no more than one DLT occurred in any of the explored dose levels up to 13 mg/m^2, thus, the MTD as defined by the protocol was not reached in this study.
Time Frame: Cycle 1 (21 days)
Population: Maximum tolerated dose (MTD) determining population.included all patients who completed the first treatment cycle (Cycle 1) according to protocol or discontinued due to a DLT. The first cycle data from this patient population were used to determine the MTD in the Phase I part of the study.
Measure: Number; unit: Dose Limiting Toxicity (DLT)
Groups:
- Patupilone 6.5 mg/m^2 (Phase I); Patupilone 7.0 mg/m^2 (Phase I); Patupilone 7.5 mg/m^2 (Phase I); Patupilone 8.0 mg/m^2 (Phase I); Patupilone 8.5 mg/m^2 (Phase I); Patupilone 9.0 mg/m^2 (Phase I); Patupilone 9.5 mg/m^2 (Phase I); Patupilone 10.0 mg/m^2 (Phase I); Patupilone 10.5 mg/m^2 (Phase I); Patupilone 11.0 mg/m^2 (Phase I); Patupilone 11.5 mg/m^2 (Phase I); Patupilone 12.0 mg/m^2 (Phase I); Patupilone 13.0 mg/m^2 (Phase I): Patupilone was administered as a single i.v. infusion over 5 to 10 minutes (Amendment 1) until (Amendment 2) and over 10 to 20 minutes (Amendment 2) until the completion of Phase I part of the study.
Arm/Group | Patupilone 6.5 mg/m^2 (Phase I) | Patupilone 7.0 mg/m^2 (Phase I) | Patupilone 7.5 mg/m^2 (Phase I) | Patupilone 8.0 mg/m^2 (Phase I) | Patupilone 8.5 mg/m^2 (Phase I) | Patupilone 9.0 mg/m^2 (Phase I) | Patupilone 9.5 mg/m^2 (Phase I) | Patupilone 10.0 mg/m^2 (Phase I) | Patupilone 10.5 mg/m^2 (Phase I) | Patupilone 11.0 mg/m^2 (Phase I) | Patupilone 11.5 mg/m^2 (Phase I) | Patupilone 12.0 mg/m^2 (Phase I) | Patupilone 13.0 mg/m^2 (Phase I)
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 5
Dose Limiting Toxicity (DLT)
  Asthenia | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Diarrhea | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Any DLT | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

5. Primary Outcome: Phase II: Number of Participants With Best Overall Response Rate (ORR) According to Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Overall response is the number of participants who had a complete response (CR) or a partial response (PR) based on local investigator's assessment of RECIST criteria. Per RECIST: CR, all detectable tumor has disappeared; PR, a >=30% decrease in the sum of the longest dimensions of the target lesions (TLs) taking as a reference the baseline sum, no worsening of non-TLs, and no new lesions; Progressive disease (PD), a >=20% increase in TLs, clearly worsening of non-TLs, or emergence of new lesions; Stable Disease (SD), small changes that do not meet previously given criteria.
Time Frame: At baseline, then every second cycle (approximately every 6 weeks), until disease progression or discontinuation. Average 18 weeks.
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Patupilone 10 mg/m^2 (Phase II) NSCLC Cohort
Number analyzed (Participants) | 35
Participants
  Complete Response | 0 [6.596 to 30.55]
  Partial Response (PR) | 6
  Stable Disease (SD) | 9
  Progressive Disease (PD) | 13
  Unknown | 7
  Best overall response (CR, PR) & the response rate | 6

6. Secondary Outcome: Duration of Stable Disease-Phase I and Phase II
Description: Duration of stable disease (CR, PR, or SD) by RECIST was defined as the time from start of study drug to the date of first documented disease progression or discontinuation due to disease progression, or death from underlying cancer, whichever event occured first.
Time Frame: Imaging was assessed every second cycle (i.e. approximately every 6 weeks), until disease progression or discontinuation from treatment . Average 18 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Patupilone (EPO906) Phase I | Patupilone (EPO906) Phase II
Number analyzed (Participants) | 50 | 35
Months | 3.7 [3.5 to 4.9] | 5.6 [3.5 to 9.0]

7. Secondary Outcome: Time to Overall Response -Phase I and Phase II
Description: Time to overall response (CR or PR) measured by RECIST was the time between study start until date of first documented response (CR or PR).
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Patupilone (EPO906) Phase I | Patupilone (EPO906) Phase II
Number analyzed (Participants) | 50 | 35
Months | 2.6 [1.2 to 3.5] | 3.4 [1.0 to 6.5]

8. Secondary Outcome: Duration of Overall Response -Phase I and Phase II
Description: Duration of overall response (CR or PR) measured by RECIST was measured from the first documented CR or PR to the date of first documented disease progression or discontinuation due to disease progression, or death from underlying cancer, whichever event occured first.
Time Frame: Duration of response according to RECIST from start of study until study discontinuation. Duration of response was assessed every second cycle ( i.e. approximately every 6 weeks) until disease progression or discontinuation from study. Average 18 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Patupilone (EPO906) Phase I | Patupilone (EPO906) Phase II
Number analyzed (Participants) | 50 | 35
Months | 2.6 [2.3 to 2.6] | NA [2.5 to NA] — Median duration was not calculated due to small number of participants (4). Outer bound of the 95% CI was not attained

ADVERSE EVENTS:
Groups:
- Patupilone 10 mg/m^2 (Phase II) NSCLC w. Brain Metastases (BM): Patupilone was administered as a single i.v. infusion over 20 minutes (Amendment 4), once every 3 weeks.
Arm/Group | Patupilone ≤7.0 mg/m^2 (Phase I) | Patupilone 7.5-8.0 mg/m^2 (Phase I) | Patupilone 8.5-9.5 mg/m^2 (Phase I) | Patupilone 10.0-11.5 mg/m^2 (Phase I) | Patupilone 12.0-13.0 mg/m^2 (Phase I) | Patupilone 10 mg/m^2 (Phase II) NSCLC Cohort | Patupilone 10 mg/m^2 (Phase II) NSCLC w. Brain Metastases (BM)
Serious Adverse Events (participants affected / at risk) | 3/6 | 3/12 | 2/12 | 3/12 | 4/8 | 14/35 | 2/4
Other Adverse Events (participants affected / at risk) | 6/6 | 11/12 | 12/12 | 10/12 | 8/8 | 33/35 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patupilone ≤7.0 mg/m^2 (Phase I) (N=6) | Patupilone 7.5-8.0 mg/m^2 (Phase I) (N=12) | Patupilone 8.5-9.5 mg/m^2 (Phase I) (N=12) | Patupilone 10.0-11.5 mg/m^2 (Phase I) (N=12) | Patupilone 12.0-13.0 mg/m^2 (Phase I) (N=8) | Patupilone 10 mg/m^2 (Phase II) NSCLC Cohort (N=35) | Patupilone 10 mg/m^2 (Phase II) NSCLC w. Brain Metastases (BM) (N=4)
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 1 | 8 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patupilone ≤7.0 mg/m^2 (Phase I) (N=6) | Patupilone 7.5-8.0 mg/m^2 (Phase I) (N=12) | Patupilone 8.5-9.5 mg/m^2 (Phase I) (N=12) | Patupilone 10.0-11.5 mg/m^2 (Phase I) (N=12) | Patupilone 12.0-13.0 mg/m^2 (Phase I) (N=8) | Patupilone 10 mg/m^2 (Phase II) NSCLC Cohort (N=35) | Patupilone 10 mg/m^2 (Phase II) NSCLC w. Brain Metastases (BM) (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 4 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Scotoma (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 4 | 2 | 2 | 3 | 0 | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 5 | 3 | 4 | 0 | 10 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 1 | 1 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 3 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 6 | 9 | 7 | 7 | 29 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 3 | 4 | 5 | 3 | 6 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 4 | 5 | 3 | 3 | 12 | 1
Asthenia (General disorders) | 1 | 2 | 3 | 0 | 1 | 11 | 0
Axillary pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 2 | 3 | 3 | 3 | 0
Face oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 2 | 4 | 3 | 3 | 5 | 1
Feeling hot (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 3 | 3 | 1 | 2 | 4 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood magnesium decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 5 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 1 | 1 | 8 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 1 | 0 | 4 | 12 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 5 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 3 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 1 | 0 | 3 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 6 | 0
Paraesthesia (Nervous system disorders) | 2 | 1 | 3 | 3 | 2 | 8 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Depression (Psychiatric disorders) | 1 | 0 | 2 | 1 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 1 | 8 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 5 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.